CLINICAL TRIAL: NCT06499454
Title: Adequacy Assessment of Bronchoscopic Biopsy Samples Using a Novel Instrument
Status: Not yet recruiting | Type: Observational
Sponsor: Ruby Robotics Inc (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RUBY2407
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Lung Diseases
Keywords: lung biopsy; bronchoscopy
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with suspected lung disease undergoing routine bronchoscopic biopsy
  Interventions: Diagnostic Test: Ruby ROSE evaluation

INTERVENTIONS:
Diagnostic Test: Ruby ROSE evaluation — Creation and digitization of ROSE slides produced using Ruby's instrument from bronchoscopic biopsy samples

SUMMARY:
The goal of this study is to learn whether the Ruby Robotics system enables pathologists to determine whether a bronchoscopic biopsy sample is adequate for diagnosis. The main question it aims to answer is:

- Are pathologists' evaluations of Ruby digital images concordant with their evaluations of manually created rapid on-site evaluation slides?

ELIGIBILITY:
Inclusion Criteria:

* The subject will undergo a planned, non-emergent transbronchial lung and/or thoracic lymph node biopsy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from patients undergoing routine transbronchial lung and/or thoracic lymph node biopsy procedures
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Concordance between pathologists' rapid evaluations of Ruby images and manually-prepared slides | 2 months from time of sample collection

SECONDARY OUTCOMES:
Pathologist ratings of quality metrics for Ruby images and manually-prepared slides | 2 months from time of sample collection